CLINICAL TRIAL: NCT04813029
Title: Defining High-Resolution Manometry Thresholds of Backward Pressure Across the Lower Esophageal Sphincter Through Straight Leg Raise Maneuver Predictive of Pathologic Acid Exposure Time
Brief Title: Thresholds of Straight Leg Raise Maneuver During High-Resolution-Manometry
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Milan (Other)
Collaborators: Medical University of Vienna (Other); University Hospital Padova (Other); University of Missouri, St. Louis (Other); Hospital Universiti Sains Malaysia (Other); The Oregon Clinic (Other); The Functional Gut Clinic (Other); University of Texas at Austin (Other); University of Athens (Other); Ohio State University (Other); University of Campania Luigi Vanvitelli (Other); Jikei University School of Medicine (Other)
Responsible Party: Principal Investigator, Luigi Bonavina, Professor, University of Milan
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: SLR2021
Record Dates: First submitted 2021-03-17; First posted 2021-03-24 (Actual); Last update posted 2021-07-22 (Actual); Status verified 2021-07

CONDITIONS: Gastroesophageal Reflux
Keywords: High Resolution Manometry; pH-impedance; Gastroesophageal Reflux disease
MeSH Terms: conditions — Gastroesophageal Reflux

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Straight Leg Raise (Experimental): Patients perform straight leg raise maneuver at the end of High-resolution Manometry test
  Interventions: Procedure: Straight leg raise maneuver

INTERVENTIONS:
Procedure: Straight leg raise maneuver — With the patient in supine position, one leg is raised to form an angle of at least 45 degrees with the bed. The patient will be asked to keep that position for at least 5 seconds. The maneuver will be repeated after 20-30 seconds. The first adequate maneuver will be considered for the study. Intra-esophageal and intra-abdominal pressure will be analyzed both during baseline and SLR maneuver. Intra-esophageal pressure is measured as peak and mean over 5 seconds, 1 cm and 5 cm above the proximal margin of the LES. Intra-abdominal pressure will be measured as peak and mean over 5 seconds 1 cm below the distal margin of the diaphragm notch.

SUMMARY:
High resolution manometry (HRM) is a key test in the preoperative assessment of patients with gastro-esophageal reflux disease (GERD) who are potential candidates for antireflux surgery. The recent Lyon consensus suggested the potential usefulness of HRM in diagnosing GERD, however, sensitivity and specificity of HRM for GERD remains low (53.6% and 72.5% respectively). Among recently proposed provocative tests during manometry, a traditional maneuver (straight leg raise maneuver, SLR) appeared promising in predicting reflux.

This is a multicenter study involving high-volume esophageal function laboratories around the world. Patients with suspected GERD and tested with HRM and pH-impedance will be asked to perform SLR during HRM. Intra-abdominal and intra-esophageal pressure during SLR will be recorded and compared with acid exposure time (AET) at pH-impedance.

Primary aim is to determine the optimal threshold of intra-esophageal pressure augmentation during straight leg raise (SLR) maneuver that predicts pathological esophageal acid exposure time (AET). Secondary aim is to assess the diagnostic performance of HMR with SRL maneuver, calculating sensitivity, specificity, false-positive rate (FPR), false-negative rate (FNR), positive predictive value and total misclassification rate.

DETAILED DESCRIPTION:
It has been demonstrated a low sensitivity and specificity of HRM for GERD (53.6% and 72.5% respectively), since there was a significant overlap between patients and controls in the majority of parameters. Masuda et al. attempted to improve HRM accuracy using a comprehensive index and new parameters, such as the backflow preventive and promotive pressure through the lower esophageal sphincter (LES). Although a significant correlation between reflux burden and the new index was found, sensitivity and specificity of HRM for GERD remained unchanged.

Recently, provocative tests have been added to the standard protocol of HRM studies. Among these, a traditional maneuver in water perfused manometry (straight leg raise maneuver, SLR) appeared promising in predicting reflux even with HRM.

A multicenter study with a large number of patients could provide more precise thresholds to predict pathologic esophageal acid exposure time and proof of real-life generalizability of SLR.

A thorough clinical evaluation will be performed. GerdQ, GERD Health Related Quality of Life (GERD-HRQL) and Reflux Symptom Index (RSI) questionnaires will be administered. HRM will be performed according to the standard protocol defined by Chicago Classification 4.0. Upon completion of the test, the SLR maneuver will be performed. With the patient in supine position, one leg is raised to form an angle of at least 45 degrees with the bed. The patient will be asked to keep that position for at least 5 seconds. The maneuver will be repeated after 20-30 seconds. The first adequate maneuver will be considered for the study. Intra-esophageal and intra-abdominal pressure will be analyzed both during baseline and SLR maneuver. Intra-esophageal pressure is measured as peak and mean over 5 seconds, 1 cm and 5 cm above the proximal margin of the LES. Intra-abdominal pressure will be measured as peak and mean over 5 seconds 1 cm below the distal margin of the diaphragm notch.

Primary aim is to determine the optimal threshold of intra-esophageal pressure augmentation during straight leg raise (SLR) maneuver that predicted pathological esophageal acid exposure time (AET). Secondary aim is to assess the diagnostic performance of HMR with SRL maneuver in patients with GERD symptoms, calculating sensitivity, specificity, false-positive rate (FPR), false-negative rate (FNR) and total misclassification rate.

The Principal Investigator will maintain research data on an encrypted file server with access controls only accessible to approved study investigators. Research records will be de-identified using coded subject identifiers prior to transfer from sites to the Principal Investigator to protect patient confidentiality. Study data will be maintained by the Principal Investigator and deleted 3 years after the end of the study.

Data from each site will be electronically transferred to Principal Investigator. The electronic copy will contain no patient identifying data elements such as name, date of birth, medical record numbers. Participating institutions will create unique patient participant numbers based on a standard formula allocated by Principal investigator (two digit institution code, two digit patient identifier, 01-20).

ELIGIBILITY:
Inclusion Criteria:

* Complete and adequate HRM and pH-impedance study performed within 2 weeks
* Successfully performed SLR maneuver (adequate intra-abdominal pressure augmentation)

Exclusion Criteria:

* Patients with prior foregut surgery
* Obese with BMI>35 Kg/m2
* Paraesophageal hiatal hernia
* Scleroderma
* Eosinophilic esophagitis

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 336 (Estimated)
Dates: Start 2021-06-01 (Actual); Primary Completion 2021-12-30 (Estimated); Study Completion 2021-12-30 (Estimated)

PRIMARY OUTCOMES:
Peak esophageal pressure during SLR | Through study completion, an average of 6 months
  Peak esophageal pressure during straight leg raise maneuver, measured 5 cm above the lower esophageal sphincter
Mean esophageal pressure during SLR | Through study completion, an average of 6 months
  Mean esophageal pressure during straight leg raise maneuver, measured 5 cm above the lower esophageal sphincter

CONTACTS AND LOCATIONS:
Overall Officials: Luigi Bonavina, MD, Principal Investigator — University of Milan
Locations (1):
- IRCCS Policlinico San Donato, San Donato Milanese, Milano, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rogers BD, Rengarajan A, Ali IA, Hasak SL, Hansalia V, Gyawali CP. Straight leg raise metrics on high-resolution manometry associate with esophageal reflux burden. Neurogastroenterol Motil. 2020 Dec;32(12):e13929. doi: 10.1111/nmo.13929. Epub 2020 Jul 6. PMID 32633016
- [Background] Masuda T, Mittal SK, Kovacs B, Csucska M, Bremner RM. Simple Manometric Index for Comprehensive Esophagogastric Junction Barrier Competency Against Gastroesophageal Reflux. J Am Coll Surg. 2020 May;230(5):744-755e3. doi: 10.1016/j.jamcollsurg.2020.01.034. Epub 2020 Mar 3. PMID 32142925
- [Background] Yadlapati R, Kahrilas PJ, Fox MR, Bredenoord AJ, Prakash Gyawali C, Roman S, Babaei A, Mittal RK, Rommel N, Savarino E, Sifrim D, Smout A, Vaezi MF, Zerbib F, Akiyama J, Bhatia S, Bor S, Carlson DA, Chen JW, Cisternas D, Cock C, Coss-Adame E, de Bortoli N, Defilippi C, Fass R, Ghoshal UC, Gonlachanvit S, Hani A, Hebbard GS, Wook Jung K, Katz P, Katzka DA, Khan A, Kohn GP, Lazarescu A, Lengliner J, Mittal SK, Omari T, Park MI, Penagini R, Pohl D, Richter JE, Serra J, Sweis R, Tack J, Tatum RP, Tutuian R, Vela MF, Wong RK, Wu JC, Xiao Y, Pandolfino JE. Esophageal motility disorders on high-resolution manometry: Chicago classification version 4.0(c). Neurogastroenterol Motil. 2021 Jan;33(1):e14058. doi: 10.1111/nmo.14058. PMID 33373111
- [Background] Gyawali CP, Kahrilas PJ, Savarino E, Zerbib F, Mion F, Smout AJPM, Vaezi M, Sifrim D, Fox MR, Vela MF, Tutuian R, Tack J, Bredenoord AJ, Pandolfino J, Roman S. Modern diagnosis of GERD: the Lyon Consensus. Gut. 2018 Jul;67(7):1351-1362. doi: 10.1136/gutjnl-2017-314722. Epub 2018 Feb 3. PMID 29437910
- [Background] van Hoeij FB, Smout AJ, Bredenoord AJ. Predictive value of routine esophageal high-resolution manometry for gastro-esophageal reflux disease. Neurogastroenterol Motil. 2015 Jul;27(7):963-70. doi: 10.1111/nmo.12570. Epub 2015 Apr 30. PMID 25930019
- [Derived] Siboni S, Kristo I, Rogers BD, De Bortoli N, Hobson A, Louie B, Lee YY, Tee V, Tolone S, Marabotto E, Visaggi P, Haworth J, Ivy M, Greenan G, Facchini C, Masuda T, Yano F, Perry K, Balasubramanian G, Theodorou D, Triantafyllou T, Cusmai L, Boveri S, Schoppmann SF, Gyawali CP, Bonavina L. Improving the Diagnostic Yield of High-Resolution Esophageal Manometry for GERD: The "Straight Leg-Raise" International Study. Clin Gastroenterol Hepatol. 2023 Jul;21(7):1761-1770.e1. doi: 10.1016/j.cgh.2022.10.008. Epub 2022 Oct 19. PMID 36270615